CLINICAL TRIAL: NCT05533853
Title: Different Methods of Forward Head Posture Correction: Does it Matter? A Randomized Controlled Study
Brief Title: Different Methods of Forward Head Posture Correction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Ibrahim Moustafa, Professor-chair of Physiotherapy Department, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo192022
Record Dates: First submitted 2022-09-05; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Forward Head Posture
Keywords: Forward head posture; Elderly; Randomized controlled trial

STUDY DESIGN:
Intervention Model Description: A prospective, double blinded, parallel-group, randomized clinical trial was conducted at one of our university's research departments,
Who Masked: Outcomes Assessor
Masking Description: The treating therapist, for both the control and intervention groups, was unblinded to the treatment method but the assessor who conducted the measurements were blinded. Assessor blinding was obtained through an independent research assist; not knowing the study design and not specifically involved in any aspect of the trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional exercise (Active Comparator): The exercise group will receive a posture corrective exercise program in the form of two strengthening(deep cervical flexors and shoulder retractors)and two stretching (cervical extensors and pectoral muscles) exercises. The exercise program will be done according to Harman et al.'s protocol and based on Kendall et al.'s approach.
  Interventions: Other: Posture corrective exercises
- Denneroll extension traction (Experimental): Denneroll extension traction. Participants in the intervention group will receive the Denneroll cervical orthotic . In the current study, Denneroll cervical traction will be used to restore the normal cervical alignment. . We will follow previously published protocols and procedures for application of this orthotic. The Denneroll orthotic will be performed in the physiotherapy clinic setting. The participants will be instructed to lie supine on the floor, in a straightened position, with their arms gently folded across their stomach.
  Interventions: Other: Denneroll extension traction

INTERVENTIONS:
Other: Posture corrective exercises — The exercises are of two types strengthening exercises and starching exercise ,). The strengthening exercises are to be done for 15 repetitions in 2 sets, Progression will be by increasing to 3 sets and adding 1 Kilogram of resistance in dumbbells exercises, the targeted muscles are teres minor, infraspinatus, medial and lower trapezius, rhomboids, and cervical flexor muscles. On the other hand, stretching exercises are to be hold for 30 seconds for 2 sets then progressed to 3 sets, the targeted muscles are pectoralis minor, sternocleidomastoid and levator scapulae.
  Arms: Traditional exercise
Other: Denneroll extension traction — The participants will be instructed to lie supine and keep their legs extended. Based on the apex of each participant's cervical curvature on the initial radiograph, the therapist will position the apex of the denneroll in one of two regions (mid cervical placement or lower cervical placement). The duration of the traction session will start at 2-3 min and increased 1 min per session until reaching the goal of 20 min, the traction will repeated three times per week for 6 weeks
  Arms: Denneroll extension traction

SUMMARY:
The goal of the study is to compare various methods of correcting forward head posture in elderly subjects. In particular, we will contrast two methods: the conventional program, which aims to restore muscle balance, and the Chiropractic BioPhysics (CBP) rehabilitation program, which relies on stretching the viscous and plastic elements of the longitudinal ligament and intervertebral disc in addition to effectively stretching the soft tissue throughout the entire body.

DETAILED DESCRIPTION:
Forward head posture has been shown to be a common postural displacement, with a conservative estimate being 66% of the whole population. It is generally believed that this abnormal posture is associated with the development and persistence of many disorders. There are many strategies to treat forward head posture; the commonly used is traditional exercise program, which aims to restore muscle balance by stretching the short muscles and strengthening the weak ones. The second treatment method is Chiropractic BioPhysics (CBP) rehabilitation program which depend on stretching of the viscous and plastic elements of the longitudinal ligament and intervertebral disc, in addition to effectively stretching the soft tissue through the entire neck area in the direction of the normal head and neck postures as seen with Denneroll traction in addition to mirror image exercise. Up to our knowledge, there is no available studies evaluating the difference between the two forward head correcting methods regarding the amount of head posture correction and the impact of different correction methods on balance. Most important, in the majority of the previous studies which investigated the efficacy of the different posture correction techniques, the subjects were young people. Therefore, the results might not be applicable to all age groups, particularly to the elderly, due to age-related musculoskeletal and physiological changes. Accordingly, the aim of this study is to compare between traditional exercise program and chiropractic biophysics approach in elderly subject .

ELIGIBILITY:
Inclusion Criteria:

* craniovertebral angle (CVA) is less than 50°

Exclusion Criteria:

* any signs or symptoms of medical "red flags" were present: tumor, fracture, rheumatoid arthritis, severe osteoporosis, and prolonged steroid use.
* Subjects with previous spine surgery
* Neurological diseases
* Vascular disorders

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-10 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
The change in craniovertebral angle | will be measured at two intervals ;pre-treatment and immediately after treatment
  The craniovertebral angle will be measured by taking a lateral photograph. The participants will be asked to sit on a chair as usual and a lateral photograph will be taken. Adhesive markers will be fixed on the tragus of the ear and the spinous processes of the seventh cervical vertebra. The head forward angle will be measured as an angle between a line drawn from the tragus of the ear to the seventh cervical vertebra and horizontal line

SECONDARY OUTCOMES:
The change in pain intensity | will be measured at two intervals ;pre-treatment and immediately after treatment
  Measurement of pain will be performed by using a visual analogue scale (VAS). The subjects will be asked about the perception of pain using a 10-cm line with 0 (no pain) on one end and 10 (worst pain) on the other. subjects will be asked to place a mark along the line to denote their level of pain
The change in Neck Disability Index | will be measured at two intervals ;pre-treatment and immediately after treatment
  The Neck Disability Index , consisting of 10 items related to daily living activities.
Changes in Cervical joint position sense testing | will be measured at two intervals ;pre-treatment and immediately after treatment
  Assessment of head repositioning accuracy with a cervical range of motion (CROM) device will be done according to existing investigations . Participants will be placed in upright neutral seated posture on a stool with no back rest with their feet touching the ground; where their perceived natural head position was determined and used as the reference neutral point. The CROM device will be positioned to 0, 0, 0 for x, y, and z rotational displacements. With their eyes closed, participants will be asked to remember their NHP as the starting posture, andthen actively rotate their head 30° to the left about the vertical y-axis and then reposition their head back the natural head position

CONTACTS AND LOCATIONS:
Locations (1):
- Ibrahim Moustafa, Sharjah city, United Arab Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No